CLINICAL TRIAL: NCT06757946
Title: Effect of Mulligan Medial/Lateral Glide With and Without Compression/ Decompression Technique on Pain, Range of Motion and Function on Patients With Knee Osteoarthritis
Brief Title: Effect of Mulligan Medial/Lateral Glide w/wo Compression/Decompression Technique on Pain ROM and Function KO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/761
Record Dates: First submitted 2024-12-26; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Combination Product: Mulligan Medial/Lateral glide with compression/ decompression technique
- Interventional group II (Active Comparator)
  Interventions: Combination Product: Mulligan Medial/Lateral glide

INTERVENTIONS:
Combination Product: Mulligan Medial/Lateral glide with compression/ decompression technique — Warm up (10 minutes with hot pack) and cool down exercises for a period of 5 to 10 minutes was given before starting and after the completion of exercises in supervised exercise program in all the groups. The following ergonomical advice were given to all the subjects, Avoid extreme knee bent positions, avoid squatting, crossed-leg sitting, frequent stair climbing or lifting heavy objects, avoid fatiguing postures except for infrequent short durations tasks, change posture frequently and use support where possible and avoid giving excess strain to the knees.
  Mulligan mobilisation consisted of Medial glide mobilisation with movement, Lateral glide mobilisation with movement, with active knee flexion (61) depending on the subjects condition. The gliding force was sustained while the patient performed 3 sets of 10 repetitions.
  Total 12 treatment sessions was given to each subject with the frequency of 3 sessions per week for 4 consecutive weeks.
  Arms: Interventional group I
Combination Product: Mulligan Medial/Lateral glide — Warm up (10 minutes with hot pack) and cool down exercises for a period of 5 to 10 minutes was given before starting and after the completion of exercises in supervised exercise program in all the groups. The following ergonomical advice were given to all the subjects, Avoid extreme knee bent positions, avoid squatting, crossed-leg sitting, frequent stair climbing or lifting heavy objects, avoid fatiguing postures except for infrequent short durations tasks, change posture frequently and use support where possible and avoid giving excess strain to the knees.
  Total 12 treatment sessions was given to each subject with the frequency of 3 sessions per week for 4 consecutive weeks. After completing the therapeutic session, post- intervention data of the outcome parameters were taken.
  Arms: Interventional group II

SUMMARY:
The Effect of Mulligan Medial/Lateral Glide Techniques with and without Compression-Decompression on Pain, Range of Motion and Function in Patients with Knee Osteoarthritis. This study aims to investigate these effects to develop more effective, non-invasive treatment protocols for improving pain, range of motion and overall function in knee OA

DETAILED DESCRIPTION:
patients, for the better understanding of response by both treatments (i.e Mulligan medial/lateral glide with and without compression/decompression technique). Patient which meet inclusion criteria, gave their consent.

ELIGIBILITY:
Inclusion Criteria

* Unilateral Knee OA, Males and females between 30 and 60 years of age,
* Patients with restricted ROM,
* Patients are having more than grade III strength of knee muscles,
* l Willingness to take part in the intervention and evaluations

Exclusion Criteria:

* Patients having unstable knee joint after Total Knee Arthroplasty or medical conditions affecting rehabilitation,
* l Joint infection of hip and knee,
* l Soft tissue injuries around knee joints,
* including tendinitis and bursitis,
* l Any fracture including patellar fracture, femur or tibia

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Pain Rating Scale (NPRS) | 12 Months
  This tool was utilized to assess the intensity of pain. A score of 0 denotes ""having no pain at all,"" while a score of 10 indicates ""the worst pain I've ever experienced."" The participants were asked to choose a number on the scale that accurately represented how much knee discomfort they were experiencing.According to a study conducted on individuals with knee OA, the interclass correlation was 0.95. Higher scores denote more intense pain; scores range from 0 to 10.
Western Ontario and McMaster Osteoarthritis Index (WOMAC) | 12 months
  It is commonly used to assess lower extremity functional status, discomfort, and associated stiffness. The questionnaire consists of twenty-four questions: seventeen pertain to physical status, five concern pain status, and two address stiffness. Each question contains five alternatives starting from 0 which signifies no symptom or trouble at all to 4 which represents considerable difficulty in doing activities with severe symptoms. There are subscale scores for stiffness, discomfort, and functional status. The sum of the 24 items that were listed, with scores ranging from 0 to 96, was the definition of the total scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Services Hospital, Shadman 1, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No